CLINICAL TRIAL: NCT07301268
Title: MC230719 Window Of Opportunity Study Of GI-102 In Patients With Recurrent High-Grade Glioblastoma
Brief Title: GI-102 Alone or With Pembrolizumab Before Surgery for Treatment of Recurrent or Progressive IDH Wildtype Glioblastoma and IDH Mutated Grade 4 Astrocytoma
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Delay in drug shipping
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MC230719; NCI-2025-09081 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 25-002007 (Other: Mayo Clinic Institutional Review Board); MC230719 (Other: Mayo Clinic)
Record Dates: First submitted 2025-12-22; First posted 2025-12-24 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Glioblastoma, IDH-Wildtype; Progressive Astrocytoma, IDH-Mutant, Grade 4; Progressive Glioblastoma; Progressive Gliosarcoma; Recurrent Astrocytoma, IDH-Mutant, Grade 4; Recurrent Glioblastoma, IDH-Wildtype; Recurrent Gliosarcoma; Resectable Astrocytoma; Resectable Glioblastoma
MeSH Terms: conditions — Glioblastoma; Astrocytoma; Gliosarcoma | interventions — Specimen Handling; Magnetic Resonance Spectroscopy; pembrolizumab; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A (GI-102, pembrolizumab) (Experimental): Patients receive GI-102 IV over 30-120 minutes on day 1 of cycle 1. Patients undergo surgery at least 14 days after cycle 1 day 1 treatment. Starting with cycle 2, patients may also receive pembrolizumab IV over 30 minutes on day 1 of each cycle. Cycles 2+ repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients may receive GI-102 for up to 2 years. Patients also undergo echocardiography or MUGA at screening, as well as blood sample collection and MRI or CT throughout the study.
  Interventions: Procedure: Biospecimen Collection; Drug: Bispecific CD80-lgG4Fc-IL-2v Fusion Protein GI-102; Procedure: Computed Tomography; Procedure: Echocardiography Test; Procedure: Magnetic Resonance Imaging; Procedure: Multigated Acquisition Scan; Biological: Pembrolizumab; Procedure: Surgical Procedure
- Group B (GI-102, pembrolizumab) (Experimental): Patients receive GI-102 IV over 30-120 minutes and pembrolizumab IV over 30 minutes on day 1 of cycle 1. Patients undergo surgery at least 14 days after cycle 1 day 1 treatment. Patients then receive GI-102 IV over 30-120 minutes and pembrolizumab IV over 30 minutes on day 1 of each cycle. Cycles 2+ repeat every 21 days for subsequent cycles in the absence of disease progression or unacceptable toxicity. Patients may receive GI-102 for up to 2 years. Patients also undergo echocardiography or MUGA at screening, as well as blood sample collection and MRI or CT throughout the study.
  Interventions: Procedure: Biospecimen Collection; Drug: Bispecific CD80-lgG4Fc-IL-2v Fusion Protein GI-102; Procedure: Computed Tomography; Procedure: Echocardiography Test; Procedure: Magnetic Resonance Imaging; Procedure: Multigated Acquisition Scan; Biological: Pembrolizumab; Procedure: Surgical Procedure

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Bispecific CD80-lgG4Fc-IL-2v Fusion Protein GI-102 — Given IV
  Other Names: GI 102; GI-102; GI102
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Echocardiography Test — Undergo echocardiography
  Other Names: EC; Echocardiography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNV Scan; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
Biological: Pembrolizumab — Given IV
  Other Names: BCD-201; GME 751; GME751; Keytruda; Lambrolizumab; MK 3475; MK-3475; MK3475; Pembrolizumab Biosimilar BCD-201; Pembrolizumab Biosimilar GME751; Pembrolizumab Biosimilar QL2107; Pembrolizumab Biosimilar RPH-075; Pembrolizumab Biosimilar SB27; QL2107; RPH 075; RPH-075; RPH075; SB 27; SB-27; SB27; SCH 900475; SCH-900475; SCH900475
Procedure: Surgical Procedure — Undergo surgery
  Other Names: Operation; Surgery; Surgery Type; Surgery, NOS; Surgical; Surgical Intervention; Surgical Interventions; Surgical Procedures; Type of Surgery

SUMMARY:
This phase II trial compares the effect of GI-102 alone and in combination with pembrolizumab given before surgery in treating patients with IDH wildtype glioblastoma and IDH mutated grade 4 astrocytoma that has come back after a period of improvement (recurrent) or that is growing, spreading, or getting worse (progressive). Glioblastoma is the most common and the most aggressive primary brain tumor in adults. Current standard of care includes surgical resection, radiation and chemotherapy. Treatment is often given before surgery (neoadjuvant therapy) to shrink the tumor and make it easier to remove. Treatment with GI-102, a bispecific fusion protein, may induce changes in body's immune system and may interfere with the ability of tumor cells to grow and spread. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the tumor, and may interfere with the ability of tumor cells to grow and spread. Giving GI-102 alone and in combination with pembrolizumab between neoadjuvant therapy and surgery may be safe, tolerable, and effective in treating patients with recurrent or progressive IDH wildtype glioblastoma and IDH mutated grade 4 astrocytoma.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Disease characteristics

  * Tissue-confirmed progressive or recurrent World Health Organization (WHO) grade IV IDH wildtype glioblastoma (including molecular glioblastoma and gliosarcoma); and IDH mutated WHO grade 4 astrocytoma
  * Candidates for surgical resection
* Measurable or non-measurable disease as defined by Response Assessment in Neuro-Oncology (RANO) 2.0
* Willing to undergo clinically indicated biopsy followed by resection of high-grade glioma at Mayo Clinic in Rochester, Minnesota (MN)
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0,1, or 2 and Karnofsky performance status (KPS) ≥ 60

  * NOTE: PS must be assessed (again) ≤ 7 days prior to first dose of study drug
* Hemoglobin ≥ 9.0 g/dL (obtained ≤ 15 days prior to registration)
* Absolute neutrophil count (ANC) ≥ 1500/mm^3 (obtained ≤ 15 days prior to registration)
* Platelet count ≥ 100,000/mm^3 (obtained ≤ 15 days prior to registration)
* Creatinine ≤ 1.5 x upper limit of normal (ULN) OR measured or calculated creatinine clearance (per institutional standard) must be ≥ 45 ml/min (obtained ≤ 15 days prior to registration)
* Total bilirubin ≤ 1.5 x ULN OR direct bilirubin ≤ ULN for patients with total bilirubin levels > 1.5 x ULN (obtained ≤ 15 days prior to registration)
* Aspartate transaminase (AST) AND alanine transaminase (ALT) ≤ 2.5 x ULN (obtained ≤ 15 days prior to registration)
* Amylase and lipase ≤ ULN (obtained ≤ 15 days prior to registration)
* Left ventricular ejection fraction (LVEF) ≥ 50% (obtained ≤ 29 days prior to registration)
* Negative pregnancy test done ≤ 8 days prior to registration, for persons of childbearing potential only
* Persons of childbearing potential (POCBP) or able to father a child must be willing to use adequate contraception starting with first dose through 180 days after last dose
* Provide written informed consent
* Willingness to provide blood specimens for correlative research
* Willingness to provide tissue specimens for correlative research
* Willingness to provide written informed consent for the neuro-oncology biorepository (IRB 12-003458) for archiving of tissue, cerebrospinal fluid (CSF), and/or blood samples collected on this protocol
* Willingness to return to enrolling institution for follow-up (during the active monitoring phase of the study)

Exclusion Criteria:

* Any of the following because this study involves an investigational agent, the genotoxic, mutagenic, and teratogenic effects of which on the developing fetus and newborn are unknown:

  * Pregnant persons
  * Nursing persons
  * Persons of childbearing potential or able to father a child who are unwilling to employ adequate contraception
* Signs or symptoms of life-threatening raised intracranial pressure: as determined by the treating neurosurgeon, including severe headache, nausea, decreasing level of consciousness, precluding 4-7-day delay in scheduling neurosurgery (i.e., immediate surgery is indicated, and patient cannot wait)
* Prior treatment

  * Received bevacizumab (AVASTIN) < 30 days prior to registration

    * NOTE: Bevacizumab is allowed for symptom control during the adjuvant phase of the study
  * Increasing dexamethasone dose prior to registration

    * NOTE: Patients currently on dexamethasone must be on dose ≤ 4 mg/day at time of registration
  * Received chemotherapy < 30 days prior to registration
  * Received a live vaccine < 30 days prior to registration
* Failure to recover from any adverse events related to any of the following therapies received prior to registration:

  * Major surgery < 28 days prior to registration
  * Radiation therapy < 14 days prior to registration
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Uncontrolled intercurrent illness including, but not limited to:

  * Ongoing or active infection requiring IV antibiotics
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Or psychiatric illness/social situations (e.g., drug addiction) that would limit compliance with study requirements
* Receiving any other investigational agent at the time of registration
* History of myocardial infarction ≤ 6 months, or congestive heart failure requiring use of ongoing maintenance therapy for life-threatening ventricular arrhythmias
* Active autoimmune disease that has required systemic treatment (i.e., with use of disease modifying agents, corticosteroids, or immunosuppressive drugs) ≤ 2 years prior to registration

  * NOTE: Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Concurrent known active hepatitis B (i.e., known positive hepatitis B virus [HBV] surface antigen [HBsAg] reactive) AND known active hepatitis C (i.e., hepatitis C virus [HCV] ribonucleic acid [RNA] [qualitative] detected by polymerase chain reaction [PCR]). Note: No testing for hepatitis B and hepatitis C is required unless mandated by local health authority

  * NOTE: Patients with known hepatitis B OR hepatitis C may be enrolled if they meet the following criteria:

    * Hepatitis B: Patients who are HBsAG positive are eligible if they have received HBV antiviral therapy for at least 4 weeks and have undetectable HBV viral load prior to randomization. Patients should remain on anti-viral therapy throughout the treatment phase of the trial and should follow local guidelines for HBV anti-viral therapy after completing study treatment
    * Hepatitis C: Patients with history of hepatitis C infection are eligible if HCV viral load is undetectable at screening. Patients must have completed curative anti-viral therapy at least 4 weeks prior to registration
* Known history of active TB (Bacillus tuberculosis)
* History of (non-infectious) pneumonitis or interstitial lung disease that required steroids, or current pneumonitis or interstitial lung disease
* Hypersensitivity to pembrolizumab, IL-2, GI-102 or any of its excipients
* History of allogeneic tissue/solid organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2026-01-29 (Actual); Primary Completion 2029-01-31 (Estimated); Study Completion 2034-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in pharmacodynamic markers of interest in tumor tissue | Up to 2 years
  Focused on an increase in CD8 T cell infiltration as well as a decrease in regulatory T cells in the tumor microenvironment (TME). Samples from stereotactic needle biopsy (pre-treatment) and resection (post-treatment) will be compared. For analyses looking at changes in measures before vs. after treatment, a paired sample t-test (or nonparametric Wilcoxon signed rank test if not sufficiently normally distributed) will have 80% power to detect an effect size of d = 0.675 within a treatment group (i.e. n=15 patients), and using a one-sided α of 0.05. Our utilization of a one-sided test in this setting is based on the fact that for changes before vs. after treatment, we are specifically focused on targeting an increase in CD8 T cell infiltration as well as a decrease in regulatory T cells in the TME.

SECONDARY OUTCOMES:
Overall survival (OS) | Up to 5 years
  Defined as the time from date of treatment start to date of death from any cause
Incidence of adverse events (AEs) | Up to 90 days after last dose of study treatment (an average of 2 years)
  Assessed using Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Will be evaluated and summarized based on the maximum grade for each type of AE reported along with the perceived attribution of the AE to the study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jian L Campian, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials